CLINICAL TRIAL: NCT05762770
Title: A Randomised Controlled Trial to Explore the Effect of Physiological Intracytoplasmic Sperm Injection (PICSI) on Miscarriage Rates in Assisted Conception
Brief Title: A Trial of Sperm Injection (PICSI) on Miscarriage Rates in Assisted Conception
Acronym: PICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shrewsbury and Telford Hospitals NHS Trust (Other)
Collaborators: The Shropshire and Mid Wales Fertility Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46341
Record Dates: First submitted 2023-02-07; First posted 2023-03-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Infertility; Miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard ICSI (No Intervention): Only spermatozoa with a moving tail but no forward motion will be selected for use in ICSI.
- PICSI (intervention) (Experimental): Using HA-binding as a sperm selection tool, the intervention group will have sperm selected physiologically prior to ICSI using PICSI dishes, following ORIGIO recommended methods (CooperSurgical, 2021).
  Interventions: Procedure: PICSI

INTERVENTIONS:
Procedure: PICSI — Using HA-binding as a sperm selection tool, the intervention group will have sperm selected physiologically prior to ICSI using PICSI dishes, following ORIGIO recommended methods (CooperSurgical, 2021).
  Arms: PICSI (intervention)

SUMMARY:
Physiological intracytoplasmic sperm injection (PICSI) is a technique used to select healthy, mature sperm for use in infertility treatment based on their physiological ability to bind to hyaluronan (HA), a natural compound found in the body. The relationship between sperm and hyaluronan can be used a marker of sperm maturity and optimal fertilising potential; this principle can be observed in vitro using a PICSI sperm selection device. The PICSI Dish contains microdots of hyaluronan, which only mature sperm bind to and these are selected by the embryologist prior to use in the intracytoplasmic sperm injection (ICSI) procedure. Recurrent miscarriages following infertility treatment are mainly idiopathic, but can be linked with increased chromosomal abnormalities. PICSI has been shown to result in better embryo development and reduced chromosomal abnormalities, due to selection of mature sperm with low DNA damage. Therefore, PICSI may be a useful tool for reducing the rate of miscarriage following infertility treatment.

The recent HABSelect study investigated treatment outcomes following PICSI, and whilst they concluded no effect on livebirth rate, they found a significant association in their secondary analysis between PICSI and reduced miscarriage rate compared to ICSI. The implications of the HABSelect study deserve to be explored further with miscarriage rate assessed as a primary outcome measure. This proof-of-concept randomised-controlled-trial aims to investigate whether PICSI shows some promise that would merit evaluation in a fully-powered trial to assess its efficacy as an advanced sperm selection method for the reduction of miscarriage rate. Eligible study participants will be patients undergoing fertility treatment using ICSI, who have provided consent for PICSI. Patients will be randomly allocated to two groups: the control group will receive ICSI according to standard protocol, and the intervention group will have additional sperm selection by HA-binding in a PICSI dish.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1 Background Physiological intracytoplasmic sperm injection (PICSI) is a technique used to select healthy, mature sperm for use in infertility treatment based on their physiological ability to bind to hyaluronic acid (HA), a natural compound found in the body. The relationship between sperm and HA can be used as a marker of sperm maturity and fertilising potential; this principle can be observed in vitro using a PICSI sperm selection device. The PICSI Dish contains microdots of hyaluronan, which only mature sperm bind to and these are selected by the embryologist prior to use in the intracytoplasmic sperm injection (ICSI) procedure.

   The recent HABSelect study investigated treatment outcomes following PICSI, and whilst they concluded no effect on livebirth rate, they found a significant association in their secondary analysis between PICSI and reduced miscarriage rate compared to ICSI . The implications of the HABSelect study deserve to be explored further with miscarriage rate assessed as a primary outcome measure.

   This proof-of-concept randomised-controlled-trial aims to investigate whether PICSI shows some promise that would merit evaluation in a fully-powered trial to assess its efficacy as an advanced sperm selection method for the reduction of miscarriage rate. Eligible study participants will be patients undergoing fertility treatment using ICSI, who have provided consent for PICSI. Patients will be randomly allocated to two groups: the control group will receive ICSI according to standard protocol, and the intervention group will have additional sperm selection by HA-binding in a PICSI dish.

   1.2 Rationale Advanced sperm selection techniques have been developed to improve ART outcomes to select the healthiest, mature and structurally sound sperm. It is crucial that the best sperm are selected for ICSI, yet conventional sperm preparation methods, including density gradients, swim-up, and simple wash, are limited in their capacity to select for spermatozoa with maturity and reduced DNA fragmentation.

   Recurrent miscarriages following infertility treatment are mainly resulting from unknown causes, but can be linked with increased chromosomal abnormalities from aneuploid embryos . Physiological Intracytoplasmic Sperm Injection (PICSI) is an advanced sperm selection method that selects for mature sperm with low DNA damage prior to injecting the oocytes in the ICSI procedure. PICSI has been shown to result in better embryo development and reduced chromosomal abnormalities. PICSI may be a useful tool for reducing the rate of miscarriage following infertility treatment.

   In the United Kingdom, there are restrictive policies set out by NHS clinical commissioning groups (CCGs) about access to assisted reproductive techniques, where only a limited number of IVF cycles are funded, so it is exceptionally important to maximise chances of transferring a viable embryo which will lead to a successful live birth.

   The SMWFC has a KPI target of <20% for miscarriage rate and alas the current figure for miscarriages following ICSI treatment is 24%, which is above this threshold. The purpose of this study is to investigate whether it is worth doing a larger study of efficacy to establish whether PICSI reduces the miscarriage rate and could therefore be introduced into practice.
2. STUDY OBJECTIVES

   2.1 Primary Objective To establish whether there is any promise of an effect of Physiological Intracytoplasmic Sperm Injection (PICSI) on miscarriage rate compared with conventional ICSI.

   2.2 Secondary Objective To investigate whether there is any promise of effect of Physiological Intracytoplasmic Sperm Injection (PICSI) on the fertilisation rate, embryo quality and development, clinical pregnancy rate, or implantation rate compared with conventional ICSI.

   2.3 Primary endpoint/outcome The primary outcome measure is miscarriage rate, meaning the number of pregnancy losses following biochemical pregnancy (detection of urinary hcGH). The primary outcome data collected is quantitative categorical data and analysed in a statistical Fisher's exact test.

   2.4 Secondary endpoint/outcome

   Secondary outcomes that will be compared for PICSI and ICSI:
   * Fertilisation rate, defined as the number of 2PNs per oocyte inseminated/injected.
   * Embryo development and quality assessed on day two and three in terms of morphology of embryos, degree of fragmentation, presence of vacuoles, symmetrical size of blastomeres.
   * Blastocyst development and quality assessed on day 5 and 6 according to the Gardner and Schoolcraft scoring system.
   * Implantation rate, defined as the number of fetal heartbeats or gestational sacs observed at 6-7 weeks gestation divided by the number of embryos transferred.
   * Biochemical pregnancy rate, indicated by the detection of urinary hcGH.
   * Clinical pregnancy rate based on the detection of a fetal heartbeat or the presence of fetal sac at 6-7 weeks gestation.
   * Live birth rate, as the number of live births at ≥37 weeks gestation per embryo transfer.
3. STUDY DESIGN The study will be carried out as a pilot randomised-controlled-trial, whereby patients will be randomly allocated to either the intervention (PICSI) group or control (ICSI) group. The simple randomisation aims to eliminate any bias and allows a true comparison of the groups with the additional step of physiological sperm selection in PICSI being the differing factor.

   Null hypothesis:

   There is no association between PICSI and reduced miscarriage rate compared to ICSI at the Shropshire and Mid Wales Fertility Centre.

   Study design:

   The study is a prospective randomised-controlled trial designed to compare PICSI (intervention) and standard ICSI (control). The ICSI group is suitable as a control in this study so the only differing variable is the sperm selection by HA-binding.

   Couples will be randomly assigned to receive treatment with standard ICSI or receive additional PICSI. Using HA-binding as a sperm selection tool, the intervention group will have sperm selected physiologically prior to ICSI using PICSI dishes, following ORIGIO recommended methods . Only spermatozoa with a moving tail but no forward motion will be selected for use in ICSI. The fertilisation rate, embryo development, implantation rate, clinical pregnancy rate, miscarriage rate and live birth rate will be compared between the two procedures.

   Researcher bias:

   The research student will be unblinded to the allocation of patients to treatment groups, however, treatments will be performed by independent staff who are trained ICSI practitioners.

   Sample size:

   The total sample size will be 140. The population being investigated will be couples undergoing infertility treatment with ICSI at the Shropshire and Mid-Wales Fertility Centre in Shrewsbury.

   Recruitment of participants will occur over 6 months and based on this time constraint we expect to attain 140 participants. This sample size is estimated to be appropriate for this small-scale study and feasible based on the number of ICSI treatments performed at the Shropshire and Mid-Wales Fertility Centre.
4. STUDY SETTING This is a single centre study, carried out at the Shropshire and Mid-Wales Fertility Centre, which is licensed and monitored by the Human Fertilisation and Embryology Authority. The patient recruitment and study conduct will take place at the Shropshire and Mid-Wales Fertility Centre. The patient population of interest are couples undergoing fertility treatment using ICSI at the Shropshire and Mid-Wales Fertility Centre, which is a tertiary care setting. Eligible participants will be patients coming through for treatment and will be identified by clinical staff at the centre who have access to the 'upcoming treatments' schedule.

The PICSI and ICSI procedures will take place in the embryology laboratory by qualified embryologists who are also experienced ICSI practitioners. Data collection will take place at the Shropshire and Mid-Wales Fertility Centre on password-protected secure desktop computers within a treatment database file. Processing and data analysis will be carried out using the anonymised data on the secure NHS OneDrive system.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ICSI as part of their treatment at the Shropshire and Mid-Wales Fertility Centre
* A total of 140 couples coming through for treatment who have consented to the use of
* PICSI in their treatment and participation in the PICSI study
* Both parties providing gametes for use in treatment must give consent to participate in the study

Exclusion Criteria:

• If testicular or frozen sperm samples are needing to be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Miscarriage rate | ≥37 weeks
  The primary outcome measure is miscarriage rate, meaning the number of pregnancy losses following biochemical pregnancy (detection of urinary hcGH).

SECONDARY OUTCOMES:
Fertilisation rates | ≥37 weeks
  Defined as the number of 2PNs per oocyte inseminated/injected.
Embryo development and quality | two and three days
  assessed on day two and three in terms of morphology of embryos, degree of fragmentation, presence of vacuoles, symmetrical size of blastomeres.
Blastocyst development and quality | 5 and 6 days
  Assessed on day 5 and 6 according to the Gardner and Schoolcraft scoring system.
Implantation rate | 6-7 weeks
  defined as the number of fetal heartbeats or gestational sacs observed at 6-7 weeks gestation divided by the number of embryos transferred.
Biochemical pregnancy rate | 6-7 weeks
  Indicated by the detection of urinary hcGH.
  • Clinical pregnancy rate based on the detection of a fetal heartbeat or the presence of fetal sac at 6-7 weeks gestation.
Live birth rate | ≥37 weeks
  As the number of live births at ≥37 weeks gestation per embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Jason Kasrie, MSc, ANSHCS, FIBMS,, Study Director — Shrewsbury & Telford Hospital Trust
Locations (1):
- The Shropshire and Mid-Wales Fertility Centre, Shrewsbury, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McDowell S, Kroon B, Ford E, Hook Y, Glujovsky D, Yazdani A. Advanced sperm selection techniques for assisted reproduction. Cochrane Database Syst Rev. 2014 Oct 28;(10):CD010461. doi: 10.1002/14651858.CD010461.pub2. PMID 25348679
- [Result] Lepine S, McDowell S, Searle LM, Kroon B, Glujovsky D, Yazdani A. Advanced sperm selection techniques for assisted reproduction. Cochrane Database Syst Rev. 2019 Jul 30;7(7):CD010461. doi: 10.1002/14651858.CD010461.pub3. PMID 31425620
- [Result] Hodes-Wertz B, Grifo J, Ghadir S, Kaplan B, Laskin CA, Glassner M, Munne S. Idiopathic recurrent miscarriage is caused mostly by aneuploid embryos. Fertil Steril. 2012 Sep;98(3):675-80. doi: 10.1016/j.fertnstert.2012.05.025. Epub 2012 Jun 7. PMID 22683012